CLINICAL TRIAL: NCT06207812
Title: Long-term Outcomes Associated With Juvenile-onset Mycosis Fungoides and Lymphomatoid Papulosis
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0745; NCI-2024-00109 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Lymphomatoid Papulosis; Mycosis Fungoides
MeSH Terms: conditions — Lymphomatoid Papulosis; Mycosis Fungoides

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To follow up with all our participants with juvenile-onset mycosis fungoides, check on their status, and ask them or their parents about long term outcomes associated with their condition.

DETAILED DESCRIPTION:
Primary Objective -To characterize the long-term outcomes associated with juvenile-onset mycosis fungoides (jMF) and lymphomatoid papulosis (lyp). The study will consider metrics such as 5-year and 10-year overall survival, and overall disease activity.

Secondary objective

-To characterize treatments and associated comorbidities.

ELIGIBILITY:
Inclusion Criteria:

-To be eligible, participants had to be diagnosed with jMF or lyp before age 20. In the case of participants below the age of 18, parents and not the children will be contacted for participation (children are exempt from participation as their parents may answer our study questions).

Exclusion Criteria:

-Participants older than 20 years of age at diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with juvenile-onset mycosis fungoides
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2028-01-12 (Estimated); Study Completion 2028-01-12 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Dai, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org